CLINICAL TRIAL: NCT05165095
Title: Clinical Assessment of Essential Remote Monitoring Functions in Pacemakers
Acronym: CALLIOPE
Status: Recruiting | Type: Observational
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Other Study IDs: IPBI01 - CALLIOPE
Record Dates: First submitted 2021-11-23; First posted 2021-12-21 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Bradycardia; Remote Monitoring
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Pacemaker implantation — De novo implantation, device upgrade to dual chamber or device replacement

SUMMARY:
The purpose of the clinical investigation is to document the safety and the performances of the remote monitoring functions of the ALIZEA, BOREA and CELEA pacemakers, i.e. the RAAT, the RVAT and the remote alerts.

DETAILED DESCRIPTION:
All patients will be included just after implantation and will then be followed during 48 months after inclusion.

At each on-site or remote follow-up visit (1 to 3 months, 6, 12, 24 and 48 months), performances of the remote monitoring functions and the cardiac pacing system itself will be measured, and safety will be monitored during the whole clinical investigation duration.

ELIGIBILITY:
Inclusion Criteria:

1. Patient implanted according to the most recent guidelines from the ESC, for 20 days or less (de novo implantation, device upgrade to dual chamber or device replacement)
2. Patient implanted with an ALIZEA, BOREA or CELEA dual chamber pacemaker from MicroPort CRM
3. Patient implanted with any active or passive CE marked bipolar RA lead, and any active or passive CE marked bipolar RV lead
4. Patient's pacemaker with the remote monitoring functions (i.e. the RAAT, the RVAT and the remote alerts) accepted by the patient and planned to be activated
5. Patient reviewed, signed and dated the ICF

Exclusion Criteria:

1. Patient with an elevated RV pacing threshold (strictly above 2.0 V for a pulse width of 0.5 ms or below)
2. Patient with permanent AF
3. Patient already enrolled in another clinical investigation that could confound the results of this clinical investigation (e.g., clinical investigations involving intra-cardiac device)
4. Patient implanted despite a contraindication for cardiac pacing system implantation (i.e. patient implanted with a defibrillator, patient contraindicated for a single dose of 310 μg of dexamethasone sodium phosphate, patient implanted with a tricuspid replacement heart valve or with a significant tricuspid valve disease that may lead to future replacement heart valve surgery)
5. Minor age patient (i.e. under 18 years of age)
6. Incapacitated patient, under guardianship, kept in detention, refusing to cooperate or not able to understand the purpose of this clinical investigation
7. Patient unavailable for the follow-up visits scheduled
8. Non-menopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated (class I or II) for a dual chamber pacemaker (de novo implantation, device upgrade to dual chamber or device replacement), according to the most recent guidelines from the ESC.
Sampling Method: Probability Sample
Enrollment: 206 (Estimated)
Dates: Start 2022-03-25 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Right Atrial Autothreshold values at the inclusion and the M1-M3 visits | 1 to 3 months post-inclusion visit (M1-M3)
In-clinic Right Ventricular pacing threshold values from Right Ventricular Autothreshold function at the inclusion and the M1-M3 visits | 1 to 3 months post-inclusion visit (M1-M3)
Technical remote alerts documented at the M1-M3 visit | 1 to 3 months post-inclusion visit (M1-M3)

SECONDARY OUTCOMES:
Right Atrial Autothreshold values up to the M48 visit | 48 months post-inclusion visit (M48)
In-clinic Right Ventricular pacing threshold values from Right Ventricular Autothreshold function up to the M48 visit | 48 months post-inclusion visit (M48)
Technical remote alerts documented up to the M48 visit | 48 months post-inclusion visit (M48)
Right Ventricular Autothreshold values up to the M48 visit | 48 months post-inclusion visit (M48)
Safety of ALIZEA, BOREA and CELEA pacemaker and of SMARTVIEW CONNECT remote monitoring systems up to the M48 visit | 48 months post-inclusion visit (M48)
Electrical performances (pacing thresholds, impedance & minimum sensed amplitude) of ALIZEA, BOREA and CELEA pacemaker systems up to the M48 visit | 48 months post-inclusion visit (M48)
Usability of ALIZEA, BOREA and CELEA pacemaker and of SMARTVIEW CONNECT remote monitoring systems up to the M48 visit | 48 months post-inclusion visit (M48)

CONTACTS AND LOCATIONS:
Locations (19):
- Austria (2):
  - Universitätsklinikum Krems, Krems
  - Allgemeines Krankenhaus Wien, Vienna
- Clinique Saint Joseph, Arlon, Belgium
- France (6):
  - CHU Bordeaux, Bordeaux
  - CH Chartres, Le Coudray
  - CHU Hôpital de la Timone, Marseille
  - CHU Nantes, Nantes
  - Clinique Pasteur Toulouse, Toulouse
  - CH Valence, Valence
- Germany (3):
  - Cardiologicum Hamburg, Hamburg
  - Cardiologicum Pirna, Pirna
  - Kardiologische Praxis Dr. Trautwein & Dr. Placke, Rostock
- Ziekenhuis VieCuri Venlo, Venlo, Netherlands
- Hospital Professor Doutor Fernando Fonseca, Amadora, Portugal
- Spain (2):
  - Hospital Arquitecto Marcide, Ferrol
  - Hospital Universitario Puerta de Hierro, Majadahonda
- United Kingdom (3):
  - Basildon University Hospital, Basildon
  - Kingston Hospital, London
  - Southend University Hospital, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: No